CLINICAL TRIAL: NCT04215822
Title: PHF19 Gene Expression and EZH2 Gene Deletion as Potential Biomarkers of Acute Myeloid Leukemia
Brief Title: PHF19 Gene Expression and EZH2 Gene Deletion in Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safia Abd El Hakeem Hussien abd el rahman, Assistant Lecturer, Assiut University
Other Study IDs: PHF19 and EZH2 genes in AML
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytogenetic Analysis; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — peripheral blood and bone marrrow aspirate samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute myeloid leukemia patients - control group: acute myeloid leukemia
  Interventions: Diagnostic Test: Cytogenetic analysis (FISH) for EZH2 gene deletion. -Real time PCR for PHF 19 gene expression.

INTERVENTIONS:
Diagnostic Test: Cytogenetic analysis (FISH) for EZH2 gene deletion. -Real time PCR for PHF 19 gene expression. — Cytogenetic analysis (FISH) for EZH2 gene deletion. -Real time PCR for PHF 19 gene expression.

SUMMARY:
The study aims to detect pattern of expression of PHF19 gene and EZH2 gene deletion in acute myeloid leukemia patients and detect their prognostic role on patients outcome.

DETAILED DESCRIPTION:
Acute Myeloid Leukemia (AML) is a heterogeneous clonal disorder characterized by immature myeloid cell proliferation and bone marrow failure. Diagnosis of AML is based on morphological diagnosis with proliferation of blast cells ≥ 20% of bone marrow cells, flow cytometric analysis and cytogenetic abnormalities.

The etiological agent and pathogenesis of AML are not entirely clear, only few AML cases can be accurately classified through traditional cellular morphological classification Thus, it is very difficult to judge the disease condition and predict prognosis. Improper expression of specific genes is a common finding in AML and may induce clinically relevant biological subsets. Cytogenetic abnormalities and molecular alterations provide the most powerful prognostic information in AML. Consequently, identification of novel biomarkers which could predict outcome or guide treatment choice will make more contribution to the clinical management of AML.

Gene repression is the deactivation of an active gene that causes shut down of transcription and it represents a powerful tool in controlling gene expression in order to prevent the metabolic dysregulation during the development or the differentiation program Polycomb repressive complex 2 (PRC2) is the sole enzymatic complex capable of establishing gene-repression through high-degree methylation of histone H3 at lysine 27 (H3K27), therefore it plays critical roles in regulation of normal hematopoiesis. Enhancer of Zeste Homolog 2 (EZH2) gene is the catalytic subunit of PRC2, located on chromosome 7q36.1. EZH2 gene encode EZH2 methyltransferase which mediates transcriptional inactivation through trimethylation of lysine 27 of histone H3 (H3K27me3). Methylation activity of EZH2 facilitate heterochromatin formation thereby silences gene function which is important for development, differentiation, and cell fate determination.

Accumulating studies have proved that EZH2 dysregulation is involved in human cancers. EZH2 may have a dual role in cancer development, acting as a tumour suppressor or an oncogene depending on the type of cancer. Overexpression of EZH2 was observed in numerous solid tumours, and targeting EZH2 can cause regression of carcinogenesis.

EZH2 inactivation medicated by mutation or under-expression in myelo-dysplastic syndromes (MDS) or myeloproliferative neoplasms (MPN) can contribute to disease pathogenesis and is associated with a poor prognosis. In AML, EZH2 dysregulation caused by mutation and under-expression may act as potential biomarkers predicting prognosis and guiding the treatment choice between transplantation and chemotherapy. EZH2 was found to have tumor suppressive and oncogenic functions in different phases of AML.

However, it remains to be defined whether deregulation of various PRC2-associated partners is also involved in malignancy development.

PHF 19 (PHD finger protein 19) a polycomb-like member of PRC2 cofactors, acts as a critical mediator of tumorigenesis. PHF 19 located in chromosome 9q33.2, encodes a member of the polycomb group (PcG) of proteins that functions by maintaining repressive transcriptional states of many developmental regulatory genes.

PHF19 has been shown to be a major modulator of histone methylation thereby regulating transcriptional chromatin activity. PHF19 directly recruits the polycomb repressive complex 2 (PRC2) via binding to H3K36me3 and leads to activation of Enhancer of Zeste Homolog 2 (EZH2) as enzymatic subunit of PRC2, thereby resulting in tri-methylation of H3K27. Previous studies confirmed that PHF19 is dysregulated in several types of cancer, resulting in the derepression of PRC2 target genes and can be used as a marker of aggressive disease.

To date, there is no published data about role of both PHF19 and EZH2 in AML. So, this study was designed to explain unexplored critical oncogenic pathway of AML in which PHF19 pattern of expression and EZH2 gene deletion promote malignant progression and detect their prognostic role.

Aim of the work:

1. To detect pattern of expression of PHF19 gene by polymerase chain reaction (PCR) and EZH2 gene deletion by Fluorescence in situ Hybridization (FISH) in newly diagnosed AML patients.
2. To study the association between expression PHF19 gene and EZH2 gene deletion in AML patients.
3. Evaluation of the role of EZH2 and PHF19 genes as predictor markers of AML patient outcome.

ELIGIBILITY:
Inclusion Criteria:

Adult newly diagnosed Patients with acute myeloid leukemia (AML), who fullfill the WHO criteria.

Exclusion Criteria:

* Patients with any other type of malignant tumors.
* Therapy related AML patients.
* AML on top of myeloproliferative neoplasms or MDS.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: newly diagnosed AML patients and healthy subjects as control group.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
detection of pattern of expression of PHF19 gene and EZH2 gene deletion in newly diagnosed AML patients. | 2 years
  Cytogenetic analysis (FISH) for EZH2 gene deletion.
  -Real time PCR for PHF 19 gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Somaia Abd El Rahman, Study Director — Assiut University

REFERENCES:
- [Background] Skoda RC, Schwaller J. Dual roles of EZH2 in acute myeloid leukemia. J Exp Med. 2019 Apr 1;216(4):725-727. doi: 10.1084/jem.20190250. Epub 2019 Mar 19. PMID 30890555
- [Background] Chu MQ, Zhang TJ, Xu ZJ, Gu Y, Ma JC, Zhang W, Wen XM, Lin J, Qian J, Zhou JD. EZH2 dysregulation: Potential biomarkers predicting prognosis and guiding treatment choice in acute myeloid leukaemia. J Cell Mol Med. 2020 Jan;24(2):1640-1649. doi: 10.1111/jcmm.14855. Epub 2019 Dec 3. PMID 31794134
- [Background] Ren Z, Ahn JH, Liu H, Tsai YH, Bhanu NV, Koss B, Allison DF, Ma A, Storey AJ, Wang P, Mackintosh SG, Edmondson RD, Groen RWJ, Martens AC, Garcia BA, Tackett AJ, Jin J, Cai L, Zheng D, Wang GG. PHF19 promotes multiple myeloma tumorigenicity through PRC2 activation and broad H3K27me3 domain formation. Blood. 2019 Oct 3;134(14):1176-1189. doi: 10.1182/blood.2019000578. Epub 2019 Aug 5. PMID 31383640